CLINICAL TRIAL: NCT02738242
Title: Evaluation of Usability and Human Factors in the Novus System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioness Neuromodulation (Industry)
Collaborators: Bioness Inc (Industry); Loewenstein Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Novus System Usability
Record Dates: First submitted 2016-03-03; First posted 2016-04-14 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Drop Foot; Muscle Weakness; Motor Neuron Disease, Upper
Keywords: Functional Electrical Stimulation; Upper motor neuron injury or disease; Drop foot; Thigh muscle weakness
MeSH Terms: conditions — Peroneal Neuropathies; Muscle Weakness; Motor Neuron Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Novus system users (Experimental): Sixteen (16) subjects suffering from foot drop and thigh muscles weakness due to upper motor neuron injury or disease will be recruit for this study and will receive the Novus system for daily use.
  Interventions: Device: Novus system

INTERVENTIONS:
Device: Novus system — The Novus system is a FES based neuroprosthesis, which intended to provide ankle dorsiflexion and knee flexion or extension in individuals with foot drop and thigh muscle weakness, following an upper motor neuron injury or disease.

SUMMARY:
The Novus system intended to provide ankle dorsiflexion and knee flexion or extension in individuals with foot drop and thigh muscle weakness, following an upper motor neuron injury or disease. The primary objective of the study is to evaluate the usability of the Novus system among these patients and to gain subjects' feedback regarding the device when used on a daily basis.The secondary objective is to obtain information about the performance of the system as a gait assistive device and to evaluate the subject's Quality of Life while using the system.

DETAILED DESCRIPTION:
The study will be carried out in two phases. Phase one (4 weeks) will focus on evaluating the usability of the Novus system. Phase two (8 weeks) will enable continued clinical follow up. The study will include sixteen (16) subjects suffering from foot drop and thigh muscles weakness due to upper motor neuron injury or disease; eight (8) subjects will be new users with no Functional Electrical Stimulation (FES) experience and the other eight (8) will be experienced Ness L300/Ness L300 Plus users. Phase two of the study will include only the new users.

The primary objective of the study is to evaluate the usability of the Novus system among these patients and gain subjects' feedback regarding the device when used on a daily basis. The secondary objective is to obtain information about the performance of the system as a gait assistive device and to evaluate the subject's Quality of Life while using the system. System usability will be evaluated by adapted 5 point Likert scale usability questionnaire and patient's feedback questionnaire. Quality of life (QoL) will be measured through Participation scale questionnaire and functional ambulation assessments; modified Emory Functional Ambulation Profile (mEFAP) that will be performed with and without the system and 2 minute walk test (2MWT) with and without the system.

ELIGIBILITY:
Inclusion Criteria:

* Upper motor neuron injury or disease.
* Foot drop - toe drag during walking.
* Lower limb spasticity- 0-4 according to the modified Ashworth scale.
* Responsible mental state, able to follow multiple step directions.
* Aged between 18 and 80 years old.
* At least six months post diagnosis
* Available for participating in the study.
* Able to understand and sign the informed consent form.
* Able to walk independently or with an assisting device (e.g. cane, walker etc.) / spot guarding for at least 10 meters.
* Sufficient response to electrical stimulation (visible muscle contractions in a seated or prone position of each designated muscle separately).

Exclusion Criteria:

* Subjects with a demand-type cardiac pacemaker, defibrillator or any electrical or metallic implant.
* Cancerous lesion of lower limb, present or suspected.
* Medical condition that prevents participation or would likely lead to inability to comply with the protocol [e.g.: congestive heart failure, patient receiving chemotherapy, uncontrolled epilepsy, etc.].
* Skin lesion at the site of the stimulation electrodes.
* Change in bone-joint structures of the lower limb, such as:

  * Contractures (ROM of dorsiflexion < 0)
  * Deformations; fracture or dislocation, which would be adversely affected by motion from the stimulation.
* Pregnancy.
* Diagnosis of major depression or psychotic disorder.
* Participation in another investigation that may directly or indirectly affect the study results.
* Unable to tolerate electrical stimulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire to evaluate system usability | End of week 4
  System usability will be evaluated by a usability questionnaire that was constructed according to the system's requirements. Subjects will be asked to complete a series of actions regarding the overall operation of the system. Each action will be rated in a 5 point likert scale, according to the performance. An average score will be calculated for each question.
Patients' Questionnaire to evaluate system ease of use | End of week 4
  System usability will be also evaluated by Patients' Questionnaire (section A). Subjects will be asked to provide their feedback regarding the ease of use (rated in a 5 point likert scale). An average score will be calculated for each question.

SECONDARY OUTCOMES:
Patients Questionnaire to compare quality of life with and without the Novus system. | End of week 4 and end of week 12
  Quality of Life will be evaluated by patients' questionnaire (section B). Subjects will be asked to give their feedback concerning their quality of life with and without the system after 4 weeks of use. Each question will be rated according to 5 likert scale. An average score will be calculated for each question. New users will be asked to fill in the questionnaire again, after 12 weeks of use in order to assess adaptability to the system.
Participation scale questionnaire (a sub-scale of Mayo-Portland Adaptability Inventory 4) for quality of life assessment compared to baseline | Baseline and end of week 4 and 12
  Quality of life (QoL) will be also measured through Participation scale questionnaire (a sub-scale of Mayo-Portland Adaptability Inventory 4) and will be compared to baseline results. New users will be asked to fill in the questionnaire again, after additional 8 weeks of use in order to assess changes after adaptability to the system.
Total score of modified Emory Functional Ambulation Profile (mEFAP) with the system compared to without the system. | Baseline and End of week 4
  Functional ambulation assessments will be measured through modified Emory Functional Ambulation Profile (mEFAP). The test will be performed with the system compared to without the system in order to assess orthotic effect.
Total score of modified Emory Functional Ambulation Profile (mEFAP) without the system at baseline compared to without the system after daily use with the system. | Baseline and End of week 4, 8 and 12.
  The test will be performed at baseline compared to end of week 4 after daily use with the system in order to assess therapeutic effect. New users will be also evaluated at week 8 and 12.
Walking velocity assessment using the 2 minute walk test (2MWT) with the system compared to without the system. | Baseline and End of week 4
  2 minute walk test (2MWT) will be performed with the system compared to without the system at baseline and end of week 4 in order to assess orthotic effect.
walking velocity assessment using the 2 minute walk test (2MWT) without the system at baseline compared to without the system after daily use with the system. | Baseline and End of week 4, 8 and 12.
  The test will be performed at baseline and compared to end of week 4 after daily use with the system in order to assess therapeutic effect. New users will be also evaluated at week 8 and 12.

OTHER OUTCOMES:
Number of subjects with anticipated and unanticipated adverse events | Throughout the 12 weeks of the study
  The occurence of anticipated and unanticipated events will be documented at each scheduled evaluation. In addition, subjects will be instructed to report adverse events 24 hours per day during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Sacher, MD, Principal Investigator — Lowenstain Hospital Rehabilitation Center
Locations (1):
- Lowenstain hospital rehabilitation center, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Springer S, Laufer Y, Becher M, Vatine JJ. Dual-channel functional electrical stimulation improvements in speed-based gait classifications. Clin Interv Aging. 2013;8:271-7. doi: 10.2147/CIA.S41141. Epub 2013 Feb 28. PMID 23467567
- [Background] Springer S, Vatine JJ, Lipson R, Wolf A, Laufer Y. Effects of dual-channel functional electrical stimulation on gait performance in patients with hemiparesis. ScientificWorldJournal. 2012;2012:530906. doi: 10.1100/2012/530906. Epub 2012 Oct 11. PMID 23097635
- [Background] Springer S, Khamis S, Laufer Y. Improved ankle and knee control with a dual-channel functional electrical stimulation system in chronic hemiplegia. A case report. Eur J Phys Rehabil Med. 2014 Apr;50(2):189-95. Epub 2012 Jul 23. PMID 24967447
- [Background] Yan T, Hui-Chan CW, Li LS. Functional electrical stimulation improves motor recovery of the lower extremity and walking ability of subjects with first acute stroke: a randomized placebo-controlled trial. Stroke. 2005 Jan;36(1):80-5. doi: 10.1161/01.STR.0000149623.24906.63. Epub 2004 Nov 29. PMID 15569875
- [Background] Hausdorff JM, Ring H. Effects of a new radio frequency-controlled neuroprosthesis on gait symmetry and rhythmicity in patients with chronic hemiparesis. Am J Phys Med Rehabil. 2008 Jan;87(1):4-13. doi: 10.1097/PHM.0b013e31815e6680. PMID 18158427